CLINICAL TRIAL: NCT00293059
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo- Controlled, 7 Cycle Duration (196 Days), Phase 3 Study of Oral Estradiol Valerate/Dienogest Tablets for the Treatment of Dysfunctional Uterine Bleeding.
Brief Title: Efficacy and Safety Study for the Treatment of Dysfunctional Uterine Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91469; 308960 (Other: Company internal)
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Metrorrhagia
Keywords: Dysfunctional Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Estradiol; dienogest

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027) (Experimental): A blister card consists of 28 pills taken orally once a day for 28 days (one cycle): 2 days of 3 mg estradiol valerate (EV); 5 days of 2 mg EV + 2 mg dienogest (DNG); 17 days of 2 mg EV + 3 mg DNG; 2 days of 1 mg EV; 2 days of placebo
  Interventions: Drug: Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027)
- Placebo (Placebo Comparator): Matching placebo to be taken orally daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027) — 2 days of 3 mg estradiol valerate (EV);5 days of 2 mg EV + 2 mg dienogest (DNG);17 days of 2 mg EV + 3 mg DNG;2 days of 1 mg EV;2 days of placeboA blister card consists of 28 pills taken orally once a day for 28 days (one cycle)
  Arms: Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027)
Drug: Placebo — Matching placebo to be taken orally daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the study drug is safe and effective in the treatment of dysfunctional uterine bleeding.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older
* With diagnosis of dysfunctional uterine bleeding without organic pathology
* And with at least one of the following symptoms: prolonged, frequent, or excessive bleeding

Exclusion Criteria:

* The use of steroidal oral contraceptives, or any drug that could alter oral contraception metabolism will be prohibited during the study.
* Women with history of endometrial ablation or dilatation or curettage within 2 months prior to study start will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (46):
- United States (37):
  - Women and Child, LPP, Lake Havasu City, Arizona
  - Marin Endocrine Associates, Greenbrae, California
  - Impact Clinical Trials - Los Angeles, Los Angeles, California
  - Blue Hill Medical Group, Pacific Palisades, California
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Women's Health Care, Inc., San Diego, California
  - Clinical Trial Center of Colorado, Greenwood Village, Colorado
  - Clinical Trial Center of Colorado, Littleton, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Clinical Physiology Associates, Inc., Fort Myers, Florida
  - New Age Medical Research Corp., Miami, Florida
  - Insignia Care for Women, P.A., Tampa, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Atlanta West Women's Center, Douglasville, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Physicians Research Group, Indianapolis, Indiana
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - NYU Langone Medical Center, New York, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Womens Medical Center, Bismarck, North Dakota
  - Reproductive Medical Research, Cincinnati, Ohio
  - Rapid Medical Research Inc., Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Women's Health Care Group of PA, Pottstown, Pennsylvania
  - South Carolina Clinical Research Center, Columbia, South Carolina
  - Brown Clinic, P.L.L.P., Watertown, South Dakota
  - New South Medical, Clarksville, Tennessee
  - Advanced Research Associates, Corpus Christi, Texas
  - Obstetrical & Gynecological Associates, PA, Houston, Texas
  - Research Across America, Plano, Texas
  - National Clinical Research, Inc., Richmond, Virginia
  - North Spokane Women's Clinic, Spokane, Washington
  - Dr. John Lenihan, MD, Tacoma, Washington
- Canada (9):
  - Maritimes Research Center, Bathurst, New Brunswick
  - Total Concept Health Care Inc., Kitchener, Ontario
  - Prime Health Research, Toronto, Ontario
  - Centre d'étude clinique de Montréal Inc., Montreal, Quebec
  - Les Gynecologues Associes, Montreal, Quebec
  - Clinique Recherche en Sante des Femmes Inc., Québec, Quebec
  - Clinique de Gynecologie, Shawinigan, Quebec
  - Q & T Research, Inc., Sherbrooke, Quebec
  - Clinique Médicale des Campus, Ste-Foy, Quebec

REFERENCES:
- [Result] Fraser IS, Jensen J, Schaefers M, Mellinger U, Parke S, Serrani M. Normalization of blood loss in women with heavy menstrual bleeding treated with an oral contraceptive containing estradiol valerate/dienogest. Contraception. 2012 Aug;86(2):96-101. doi: 10.1016/j.contraception.2011.11.011. Epub 2012 Jan 10. PMID 22240178
- [Result] Jensen JT, Parke S, Mellinger U, Machlitt A, Fraser IS. Effective treatment of heavy menstrual bleeding with estradiol valerate and dienogest: a randomized controlled trial. Obstet Gynecol. 2011 Apr;117(4):777-787. doi: 10.1097/AOG.0b013e3182118ac3. PMID 21422847
- [Result] Fraser IS, Parke S, Mellinger U, Machlitt A, Serrani M, Jensen J. Effective treatment of heavy and/or prolonged menstrual bleeding without organic cause: pooled analysis of two multinational, randomised, double-blind, placebo-controlled trials of oestradiol valerate and dienogest. Eur J Contracept Reprod Health Care. 2011 Aug;16(4):258-69. doi: 10.3109/13625187.2011.591456. PMID 21774563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of first participant, first visit was 14 Dec 2005. The date of last participant, last visit was 21 May 2008.
Pre-assignment Details: A total of 1077 participants were screened for inclusion into the study; 887 participants failed screening. The remaining 190 participants were randomized; 120 participants were randomized to the estradiol valerate/dienogest group and 70 participants to the placebo group.
Period: Overall Study
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Started | 120 | 70
Subjects Received Treatment | 119 | 66
Cycle 1/Treatment Day 28 | 115 | 64
Cycle 3/Treatment Day 84 | 100 | 55
Cycle 7/Treatment Day 196 | 113 (Includes participants that prematurely discontinued and may not be counted in earlier visits.) | 62 (Includes participants that prematurely discontinued and may not be counted in earlier visits.)
Completed | 85 | 51
Not Completed | 35 | 19
Not completed — Adverse Event | 12 | 4
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Pregnancy | 1 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Participant moved out of state | 1 | 0
Not completed — Participant stopped study drug | 1 | 0
Not completed — Noncompliant - sanitary pads collection | 0 | 1
Not completed — missing | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo | Total
Number analyzed (Participants) | 120 | 70 | 190
Age Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (7.5) | 37.0 (6.7) | 36.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 70 | 190
  Male | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (3.6) | 25.8 (3.6) | 26.1 (3.6)
excessive bleeding [Number; unit: participants] — 2 or more bleeding episodes in the 90-day run-in phase, each with blood loss ≥80 mL
  participants | 91 | 60 | 151
prolonged bleeding [Number; unit: participants] — 2 or more bleeding episodes in the 90-day run-in phase, each lasting 8 or more days
  participants | 26 | 12 | 38
frequent bleeding [Number; unit: participants] — > 5 bleeding episodes in the 90-day run-in phase, with a minimum of 20 bleeding days overall
  participants | 4 | 2 | 6
prolonged and frequent bleeding [Number; unit: participants] | 3 | 2 | 5
prolonged and excessive bleeding [Number; unit: participants] | 9 | 9 | 18
frequent and excessive bleeding [Number; unit: participants] | 1 | 0 | 1
prolonged, frequent and excessive bleeding [Number; unit: participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With no Dysfunctional Uterine Bleeding (DUB) Symptoms
Description: Up to 8 criteria had to be met for complete response during 90-day period. No bleeding episodes (BE) >7 days, no >4 BE, no BE with MBL >=80 mL, no >1 BE increase from baseline, no increase from baseline in an individual participant's total number of bleeding days and total number of bleeding days not >24 days. Additionally, for participants included with prolonged bleeding: decrease between maximum duration during run-in and efficacy >=2 days excessive bleeding: MBL associated with each episode decreased by >=50% from average of qualifying episodes during run-in.
Time Frame: during a time period of 90 days under treatment
Population: The intent-to-treat (ITT) group consisted of all randomized participants.
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 120 | 70
Proportion of participants | 0.292 | 0.029
Statistical Analysis 1: Comparison: Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) vs Placebo; Test type: Superiority or Other; p < 0.0001, inverting 2 one-sided tests

2. Secondary Outcome: Proportion of Participants Cured From Prolonged Bleeding
Description: Prolonged bleeding was defined as 2 or more bleeding episodes, each lasting 8 or more days in a 90-day period. Participants were considered cured if they had no bleeding episodes lasting more than 7 days and the decrease between the maximum duration during the run-in phase and the maximum duration during the efficacy phase was at least 2 days.
Time Frame: during a time period of 90 days under treatment
Population: The ITT population consisted of all randomized participants who enrolled with prolonged bleeding.
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 26 | 12
Proportion of participants | 0.154 | 0.083

3. Secondary Outcome: Proportion of Participants Cured From Frequent Bleeding
Description: Frequent bleeding was defined as greater than 5 bleeding episodes, with a minimum of 20 bleeding days overall in a 90-day period. Participants were considered cured if they had no more than 4 bleeding episodes and the total number of bleeding days did not exceed 24 days and there was no increase in the total number of bleeding days in the efficacy phase as compared to the run-in phase.
Time Frame: during a time period of 90 days under treatment
Population: The ITT population consisted of all randomized participants who enrolled with frequent bleeding.
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 4 | 2
Proportion of participants | 0.250 | 0.0

4. Secondary Outcome: Proportion of Participants Cured From Excessive Bleeding
Description: Excessive bleeding was defined as 2 or more bleeding episodes each with blood loss volume of 80 mL or more in a 90-day period. Participants were considered cured if (1) the blood loss volume associated with each episode was less than 80 mL and (2) the blood loss volume associated with each bleeding episode represented a decrease of at least 50% from the average of the qualifying bleeding episodes, where the qualifying bleeding episodes were those with a blood loss volume ≥ 80 mL (per episode) that occurred during the run-in phase.
Time Frame: during a time period of 90 days under treatment
Population: The ITT population consisted of all randomized participants who enrolled with excessive bleeding.
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 91 | 60
Proportion of participants | 0.385 | 0.05

5. Secondary Outcome: Proportion of Participants With Improvement in the Investigator's Global Assessment Scale at Treatment Day 84
Description: The investigators assessed the participants' change in DUB symptoms at day 84 (visit 7) compared with admission to the study according to a scale of 1 (very much improved) to 7 (very much worse), using the following information: central laboratory data, physical examination, e-diary data, and participant interview. Improvement was defined as being classified as a score of 3 or less.
Time Frame: from baseline up to treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 100 | 55
Proportion of participants | 0.880 | 0.509

6. Secondary Outcome: Proportion of Participants With Improvement in the Investigator's Global Assessment Scale at Treatment Day 196
Description: The investigators assessed the participants' change in DUB symptoms at day 196 (visit 11) compared with admission to the study according to a scale of 1 (very much improved) to 7 (very much worse), using the following information: central laboratory data, physical examination, e-diary data, and participant interview. Improvement was defined as being classified as a score of 3 or less.
Time Frame: from baseline up to treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 114 | 62
Proportion of participants | 0.807 | 0.419

7. Secondary Outcome: Proportion of Participants With Improvement in the Participant's Overall Assessment Scale at Treatment Day 84
Description: Participants assessed their overall improvement at day 84 (visit 7) compared with their condition at admission to the study on a scale of 1 (very much improved) to 7 (very much worse). Improvement was defined as being classified as a score of 3 or less.
Time Frame: from baseline up to treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 47
Proportion of participants | 0.835 | 0.426

8. Secondary Outcome: Proportion of Participants With Improvement in the Participant's Overall Assessment Scale at Treatment Day 196
Description: Participants assessed their overall improvement at day 196 (visit 11) compared with their condition at admission to the study on a scale of 1 (very much improved) to 7 (very much worse). Improvement was defined as being classified as a score of 3 or less.
Time Frame: from baseline up to treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 47
Proportion of participants | 0.812 | 0.383

9. Secondary Outcome: Change From Baseline in Blood Loss Volume for All Participants to the Reference Period of 90 Days Under Treatment
Description: Menstrual blood loss was determined using the alkaline hematin method for the 90 days before treatment (baseline) and for 90 days under treatment. A negative value indicates a reduction in blood loss after treatment.
Time Frame: Baseline and reference period of 90 days under treatment
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 79 | 46
mL | -353.1 (309.4) | -130.4 (338.3)

10. Secondary Outcome: Menstrual Blood Loss Volume for All Participants at Cycle 1
Description: Menstrual blood loss volume was determined using the alkaline hematin method after participants were on treatment for one cycle
Time Frame: 28 days
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 117 | 66
mL | 136.5 (141.3) | 146.9 (133.9)

11. Secondary Outcome: Menstrual Blood Loss Volume for All Participants at Cycle 3
Description: Menstrual blood loss volume was determined using the alkaline hematin method after participants were on treatment for 3 cycles
Time Frame: 28 days
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 104 | 58
mL | 59.9 (91.5) | 139.6 (92.2)

12. Secondary Outcome: Menstrual Blood Loss Volume for All Participants at Cycle 7
Description: Menstrual blood loss volume was determined using the alkaline hematin methods after participants were on treatment for 7 cycles
Time Frame: 28 days
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 86 | 49
mL | 41.3 (54.2) | 113.3 (76.6)

13. Secondary Outcome: Change From Baseline in Blood Loss Volume for Participants With Excessive Bleeding to the Reference Period of 90 Days Under Treatment
Description: The blood loss volume for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 mL or more during the run-in phase) was determined for the 90 days before treatment (ie, run-in phase) and for the 90 days under treatment. A negative value indicates a reduction in blood loss while under treatment compared to before treatment.
Time Frame: baseline and reference period of 90 days under treatment
Population: ITT, participants with excessive bleeding at baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 65 | 42
mL | -411.9 (308.5) | -152.3 (343.2)

14. Secondary Outcome: Menstrual Blood Loss Volume for Participants With Excessive Bleeding at Cycle 1
Description: The blood loss volume for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 mL or more during the run-in phase) was determined using the alkaline hematin method after participants were on treatment for one cycle.
Time Frame: 28 days
Population: ITT, participants with excessive bleeding at baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 90 | 58
mL | 206.1 (179.8) | 194.7 (132.2)

15. Secondary Outcome: Menstrual Blood Loss Volume for Participants With Excessive Bleeding at Cycle 3
Description: The blood loss volume for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 mL or more during the run-in phase) was determined using the alkaline hematin method after participants were on treatment for 3 cycles.
Time Frame: 28 days
Population: ITT, participants with excessive bleeding at baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 78 | 51
mL | 67.1 (96.2) | 147.4 (93.4)

16. Secondary Outcome: Menstrual Blood Loss Volume for Participants With Excessive Bleeding at Cycle 7
Description: The blood loss volume for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 mL or more during the run-in phase) was determined using the alkaline hematin method after participants were on treatment for 7 cycles.
Time Frame: 28 days
Population: ITT, participants with excessive bleeding at baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 68 | 42
mL | 47.5 (58.5) | 116.9 (77.5)

17. Secondary Outcome: Change From Baseline in Number of Bleeding Days to the Reference Period of 90 Days Under Treatment
Description: The number of bleeding days was determine for the 90 days before treatment (baseline) and for 90 days while under treatment. A negative value indicates a reduction in the number of bleeding days while under treatment compared to baseline.
Time Frame: baseline and reference period of 90 days under treatment
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: bleeding days
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 79 | 46
bleeding days | -5.2 (11.4) | -2.0 (6.2)

18. Secondary Outcome: Change From Baseline in Number of Bleeding Episodes to the Reference Period of 90 Days Under Treatment
Description: A bleeding episode was one that lasted for at least 2 days, and where the bleeding days were separated by no more than 1 bleeding-free day. An episode stopped with 2 consecutive bleeding-free days. The number of episodes was determined for the 90 days before treatment and for the 90 days under treatment. A negative values indicates a reduction from baseline in the number of episodes while under treatment.
Time Frame: baseline and reference period of 90 days under treatment
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: bleeding episodes
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 79 | 46
bleeding episodes | -0.5 (1.5) | -0.3 (0.9)

19. Secondary Outcome: Change From Baseline in Number of Sanitary Protection Used at 90 Days of Treatment
Description: The number of total sanitary protection items used during the 90-day run-in phase before treatment (baseline) and the number of total sanitary protection items used during the 90 days while under treatment was determined. A negative value indicates a reduction in the number of sanitary protection items used while under treatment compared to the number used before treatment.
Time Frame: baseline and reference period of 90 days under treatment
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Sanitary protection products
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 79 | 46
Sanitary protection products | -43.6 (40.9) | -21.2 (43.2)

20. Secondary Outcome: Change From Baseline in Psychological General Well-Being Index (PGWBI) Scores at Treatment Day 84
Description: The PGWBI questionnaire consisted of 22 questions that were answered using a 6-grade Likert scale. The minimum overall score was 22 and the maximum was 132. The higher the score, the better the well being of the participant. The observation phase was the last 4 weeks. The following 6 dimensions were derived from the questionnaire: anxiety, depressed mood, positive well-being, self-control, health, and vitality and the highest possible scores were 30, 18, 24, 18, 18, and 24, respectively.
Time Frame: baseline and treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 82 | 44
Scores on a scale | -1.0 (13.4) | -0.7 (10.1)

21. Secondary Outcome: Change From Baseline in Psychological General Well-Being Index (PGWBI) Scores at Treatment Day 196
Description: as for outcome 20
Time Frame: baseline and treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 81 | 43
Scores on a scale | 0.7 (14.6) | 1.0 (10.1)

22. Secondary Outcome: Change From Baseline in McCoy Female Sexuality Questionnaire (MFSQ) Scores at Treatment Day 84
Description: The MFSQ was designed to measure aspects of female sexuality and asked about the participants' sexual experience during the last 4 weeks. Higher scores represent higher, more complete, or better integrated levels of female sexual function. Minimum and maximum possible values are 19 and 133.
Time Frame: baseline and treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 42 | 22
Scores on a scale | -3.5 (12.0) | 0.8 (8.4)

23. Secondary Outcome: Change From Baseline in McCoy Female Sexuality Questionnaire (MFSQ) Scores at Treatment Day 196
Description: as for outcome 22
Time Frame: baseline and treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 37 | 24
Scores on a scale | -2.0 (15.9) | -0.8 (9.1)

24. Secondary Outcome: Change From Baseline in EuroQoL (Quality of Life) 5 Dimensional Health Questionnaire (EQ-5D) Scores at Treatment Day 84
Description: The Health State Classification of the EQ-5D comprised 5 questions addressing mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Participants were asked to indicate their current health state by ticking the most appropriate of 3 statements about each of the questions (ie, no problems, some problems, extreme problems). The best possible answers were (1,1,1,1,1), which equals a valuation score of 1.0. The worst possible answers were (3,3,3,3,3), which equals a valuation score of .594. The change from the baseline score at day 84 is presented.
Time Frame: baseline and treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 86 | 47
scores on a scale | -0.0035 (0.2145) | -0.0024 (0.1507)

25. Secondary Outcome: Change From Baseline in EuroQoL (Quality of Life) 5 Dimensional Health Questionnaire (EQ-5D) Scores at Treatment Day 196
Description: The Health State Classification of the EQ-5D comprised 5 questions addressing mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Participants were asked to indicate their current health state by ticking the most appropriate of 3 statements about each of the questions (ie, no problems, some problems, extreme problems). The best possible answers were (1,1,1,1,1), which equals a valuation score of 1.0. The worst possible answers were (3,3,3,3,3), which equals a valuation score of .594. The change from the baseline score at day 196 is presented.
Time Frame: baseline and treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 47
Scores on a scale | 0.0052 (0.1504) | 0.0154 (0.1611)

26. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) of the EQ-5D Score at Treatment Day 84
Description: The visual analogue scale (ie, "thermometer") had endpoints of 100 (best imaginable health state) at the top, and 0 (worst imaginable health state) at the bottom. Participants rated their current health state by drawing a line from the box marked 'your own health state today' to the appropriate point on the thermometer scale. The change from baseline at day 84 is presented.
Time Frame: baseline and treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 47
Scores on a scale | -2.07 (11.74) | -0.26 (10.38)

27. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) of the EQ-5D Score at Treatment Day 196
Description: The visual analogue scale (ie, "thermometer") had endpoints of 100 (best imaginable health state) at the top, and 0 (worst imaginable health state) at the bottom. Participants rated their current health state by drawing a line from the box marked 'your own health state today' to the appropriate point on the thermometer scale. The change from baseline at day 196 is presented.
Time Frame: baseline and treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 84 | 47
Scores on a scale | -0.07 (12.86) | -0.51 (12.90)

28. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Change in the Employment Status) at Treatment Day 84
Description: Participants were asked if there was any change in her employment status in the last 12 weeks. The proportion of participants with a change is displayed.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 86 | 47
Proportion of participants | 0.221 | 0.106

29. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Days Missed From Work) at Treatment Day 84
Description: Participants were asked how many days and hours they missed from work during the past 12 weeks because of problems associated with DUB, not including the time missed to participate in this study.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 75 | 41
day | 0.4 (1.84) | 0.7 (1.87)

30. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Productivity While Working) at Treatment Day 84
Description: Participants were asked to rate on a scale of 0 to 10, how much their DUB affected productivity while working during the past 12 weeks, where 0 represented that DUB had no effect on work and 10 represented that DUB completely prevented her from working.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 78 | 42
Scores on a scale | 2.38 (2.175) | 3.07 (2.088)

31. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Regular Daily Activities) at Treatment Day 84
Description: Participants were asked to rate on a scale of 0 to 10 how much DUB affected their ability to do their regular daily activities, other than work at a job, during the past 12 weeks where 0 represented that DUB had no effect on daily activities and 10 represented that DUB completely prevented her from doing daily activities.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 80 | 45
Scores on a scale | 2.81 (2.551) | 3.91 (2.466)

32. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Unscheduled Outpatient Visit at Hospital) at Treatment Day 84
Description: Participants were asked if they had any unscheduled outpatient visits to a hospital because of DUB during the past 12 weeks, not including visits that were due to participation in this study. The proportion of participants with such visits is displayed.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 86 | 47
Proportion of participants | 0.012 | 0.0

33. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Unscheduled Visit to Physician) at Treatment Day 84
Description: Participants were asked if they had any unscheduled visits to a physician (non-hospital medical care) because of DUB during the past 12 weeks, not including visits that were due to participation in this study. The proportion of participants with such visits is displayed.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 47
Proportion of participants | 0.012 | 0.0

34. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Additional Unscheduled Procedures) at Treatment Day 84
Description: Participants were asked if they had any unscheduled procedures (eg, laparoscopy, laboratory tests, ultrasound) because of DUB during the past 12 weeks. The proportion of participants with such procedures is displayed.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 86 | 47
Proportion of participants | 0.012 | 0.0

35. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Received Ambulatory Services) at Treatment Day 84
Description: Participants were asked if they had received ambulatory services (eg, home help, child care) because of DUB during the past 12 weeks. The proportion of participants who received such services is displayed.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 103 | 57
Proportion of participants | 0.0 | 0.0

36. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Out-of-pocket Expenses) at Treatment Day 84
Description: Participants were asked to specify if they had out-of-pocket expenses because of DUB during the past 12 weeks, including over-the-counter medication (the name of the medication, the number of packages, and the cost per package), co-payments due to prescribed medication, and costs to travel to and from medical appointments. The proportion of participants with such expenses is displayed.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 99 | 54
Proportion of participants | 0.323 | 0.407

37. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Any Medical Treatment) at Treatment Day 84
Description: Participants were asked if they had any medical treatment (eg, prescribed medication, other treatment) because of DUB during the past 12 weeks. The proportion of participants with such treatment is displayed.
Time Frame: treatment day 84
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 48
Proportion of participants | 0.047 | 0.062

38. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Change in the Employment Status) at Treatment Day 196
Description: Participants were asked if there was any change in employment status in the last 12 weeks. The proportion of participants with a change is displayed.
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 47
Proportion of participants | 0.129 | 0.213

39. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Days Missed From Work) at Treatment Day 196
Description: Participants were asked how many days and hours were missed from work during the past 12 weeks because of problems associated with DUB, not including the time missed to participate in this study.
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 79 | 42
days | 0.2 (1.19) | 0.4 (1.51)

40. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Productivity While Working) at Treatment Day 196
Description: Participants were asked to rate on a scale of 0 to 10, how much DUB affected their productivity while working during the past 12 weeks, where 0 represented that DUB had no effect on work and 10 represented that DUB completely prevented her from working.
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 78 | 38
Scores on a scale | 2.40 (2.293) | 4.03 (3.123)

41. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Regular Daily Activities) at Treatment Day 196
Description: Participants were asked to rate on a scale of 0 to 10 how much DUB affected their ability to do regular daily activities, other than work at a job, during the past 12 weeks where 0 represented that DUB had no effect on daily activities and 10 represented that DUB completely prevented her from doing her daily activities.
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 80 | 42
Scores on a scale | 2.48 (2.291) | 4.10 (2.903)

42. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Unscheduled Outpatient Visit at Hospital) at Treatment Day 196
Description: as for outcome 32
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 46
Proportion of participants | 0.012 | 0.0

43. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Unscheduled Visit to Physician) at Treatment Day 196
Description: as for outcome 33
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 84 | 45
Proportion of participants | 0.024 | 0.0

44. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Additional Unscheduled Procedures) at Treatment Day 196
Description: as for outcome 34
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 84 | 46
Proportion of participants | 0.024 | 0.0

45. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Received Ambulatory Services) at Treatment Day 196
Description: Participants were asked if they had received ambulatory services (eg, home help, child care) because of DUB during the past 12 weeks. The proportion of participants who had received such services is displayed.
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 81 | 45
Proportion of participants | 0.012 | 0.0

46. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Out-of-pocket Expenses) at Treatment Day 196
Description: Participants were asked to specify out-of-pocket expenses because of DUB during the past 12 weeks, including over-the-counter medication, co-payments due to prescribed medication, and costs to travel to and from medical appointments. The proportion of participants with such expenses is displayed.
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 87 | 51
Proportion of participants | 0.241 | 0.314

47. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire (Any Medical Treatment) at Treatment Day 196
Description: as for outcome 37
Time Frame: treatment day 196
Population: ITT, excluding participants with missing data
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 85 | 47
Proportion of participants | 0.047 | 0.043

48. Secondary Outcome: Change From Baseline in Hematocrit (Hct) Concentrations at Treatment Day 196
Description: Hematocrit was measured before treatment and after 196 days under treatment. A positive value indicates an increase in hematocrit from baseline at treatment day 196.
Time Frame: baseline and treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: Percentage of blood volume
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 108 | 59
Percentage of blood volume | 1.30 (2.98) | 0.09 (3.04)

49. Secondary Outcome: Change From Baseline in Serum Ferritin Concentration at Treatment Day 84
Description: Serum ferritin was measured before treatment and after 84 days under treatment. A positive value indicates an increase in serum ferritin from baseline at treatment day 84.
Time Frame: baseline and treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 99 | 54
ng/mL | 0.2 (35.6) | -1.5 (12.2)

50. Secondary Outcome: Change From Baseline in Serum Ferritin Concentration at Treatment Day 196
Description: Serum ferritin was measured before treatment and after 196 days under treatment. A positive value indicates an increase in serum ferritin from baseline at treatment day 196.
Time Frame: baseline and treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 112 | 59
ng/mL | 5.3 (37.8) | 2.0 (11.9)

51. Secondary Outcome: Change From Baseline in Hemoglobin Concentration at Treatment Day 84
Description: Hemoglobin was measured before treatment and after 84 days under treatment. A positive value indicates an increase in hemoglobin from baseline at treatment day 84.
Time Frame: baseline and treatment day 84
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 96 | 53
g/dL | 0.22 (0.83) | 0.17 (0.62)

52. Secondary Outcome: Change From Baseline in Hemoglobin Concentration at Treatment Day 196
Description: Hemoglobin was measured before treatment and after 196 days under treatment. A positive value indicates an increase in hemoglobin from baseline at treatment day 196.
Time Frame: baseline and treatment day 196
Population: ITT, excluding participants with missing data
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 108 | 59
g/dL | 0.57 (1.02) | 0.20 (1.03)

53. Post Hoc Outcome: Proportion of Participants With Successful Treatment
Description: End of Study menstrual blood loss (MBL) ≤ 80 mL and a decrease to a value of ≤ 50% of the Baseline MBL was considered as treatment success.
Time Frame: during a time period of 28 days under treatment
Population: Only participants with heavy menstrual bleeding were included in the analysis.
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 88 | 60
Proportion of participants
  End of study MBL <=80 mL | 0.568 | 0.183
  Decrease MBL >=50% of baseline MBL | 0.568 | 0.217
  Successful treatment | 0.511 | 0.133

54. Post Hoc Outcome: Change in Absolute Value From Baseline MBL to end-of Study MBL
Description: The MBL for each cycle includes intermenstrual bleeding in addition to withdrawal bleeding. Baseline MBL was the mean MBL of measured MBL during three cycles in the run-in Phase. One cycle was defined as 28 days. For this analysis, the run-in Phase was defined by the days 1 to 84 (= 3 cycles each of 28 days). End of Study MBL was measured during Cycle 7 of the Treatment Phase (data imputation and Last Observation Carried Forward was applied).
Time Frame: during a time period of 28 days under treatment
Population: Only participants with heavy menstrual bleeding were included in the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 88 | 60
mL | -114.60 (138.712) | -49.944 (117.038)

ADVERSE EVENTS:
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/119 | 2/66
Other Adverse Events (participants affected / at risk) | 46/119 | 21/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) (N=119) | Placebo (N=66)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) (N=119) | Placebo (N=66)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (9) | 5 (7)
Nasopharyngitis (Infections and infestations) | 9 (9) | 6 (7)
Vaginitis bacterial (Infections and infestations) | 7 (8) | 4 (4)
Weight increased (Investigations) | 10 (10) | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 9 (28)
Breast pain (Reproductive system and breast disorders) | 6 (8) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 6 (7) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less